CLINICAL TRIAL: NCT06903741
Title: Effect of a New Preservative-free Combination of Trehalose, Sodium Hyaluronate and N-acetyl-aspartyl-glutamate (NAAGA) on Dry Eye Disease and Patient Quality of Life
Brief Title: New Preservative-free Combination of Trehalose, Sodium Hyaluronate and N-acetyl-aspartyl-glutamate (NAAGA) in Dry Eye
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT2769-006
Record Dates: First submitted 2025-03-21; First posted 2025-04-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: T2769
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated group (Experimental): Groupe receiving T2769
  Interventions: Device: T2769

INTERVENTIONS:
Device: T2769 — Preservative-free combination of trehalose, sodium hyaluronate and N-acetyl-aspartyl-glutamate

SUMMARY:
The goal of this prospective, non-randomized, non-comparative, monocentric PMCF study is to assess the performance of a new preservative-free combination of trehalose, sodium hyaluronate and NAAGA on DED at 6 months in 30 patients having dry eye disease.

The main questions it aims to answer are:

* To assess the performance and safety of T2769 at 3 months and 6 months.
* To assess patient compliance to therapy.
* To assess the occurrence of dry eye flares. Participants will be asked to use T2769 on a daily basis and complete a self-questionnaire throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years,
* Able to give written informed consent prior the initiation of any procedure,
* History of dry eye syndrome for at least 3 months,
* OSDI ≥13,
* Never been treated with artificial tears or with no artificial tears at least 1 month before the enrolment, or not satisfied with current artificial tears.

Exclusion Criteria:

Systemic/non Ophthalmic Exclusion Criteria

* Known or suspected hypersensitivity to one of the components of the IMD,
* History of or active relevant systemic condition incompatible with the investigation or likely to interfere with the investigation results or the patient safety according to investigator judgment.

Specific Exclusion Criteria Regarding Childbearing Potential Women

* Pregnant or breast-feeding women,
* Childbearing potential women neither surgically sterilised nor using an adequate contraception (oral contraceptive, intra-uterine device, subcutaneous contraceptive implant, vaginal ring, patch) .

Exclusion Criteria Related to General Conditions

* Alcohol addiction and heavy smoker according to investigator's judgement,
* Unable to understand the investigation procedures or to give informed consent,
* Non-compliant (e.g., not willing to attend a visit or completing the self-questionnaire; way of life interfering with compliance),
* Participant in this investigation at the same time as another clinical investigation/study,
* Participant in this investigation within the exclusion period of a previous study/investigation with a minimum of one month,
* Participant being institutionalized because of legal or regulatory order, inmate of psychiatric wards, prison or state institutions, or employee or family member of the investigation sites or of the Sponsor's company.

Exclusion criteria related to previous and concomitant treatments (medications/non-medicinal therapies/procedures)

• Participant with previous, current or anticipated prohibited listed treatment (or prohibited modification of treatment regimen).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Improvement of DED signs and symptoms at 6 months (M6) according to Ocular Surface Disease Index (OSDI) score change from baseline to M6 | at baseline, at 3 months, at 6 months
  Improvement of DED signs and symptoms at 6 months (M6) according to Ocular Surface Disease Index (OSDI) score change from baseline to M6 OSDI is a 12-item scale with total score from 0 to 100 (Mild 13-22; moderate 23-32; severe 33-100)

CONTACTS AND LOCATIONS:
Locations (1):
- Group Practice Outpatient Clinic for Specialized Medical, Varna, Bulgaria